CLINICAL TRIAL: NCT02775630
Title: Assessment of the Contribution of Hypnosis in the Tolerance of the Bronchoscopy
Acronym: FIBROHYPNOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FIBRO HYPNOSE
Record Dates: First submitted 2016-05-09; First posted 2016-05-17 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Respiratory System Abnormalities
MeSH Terms: conditions — Respiratory System Abnormalities | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Examination under hypnosis in addition to local anesthesia (Experimental): Patients will have hypnosis add-on local anesthesia
  Interventions: Procedure: hypnosis
- Examination under local anesthesia (No Intervention): Patients will receive a local anesthesia only without hypnosis

INTERVENTIONS:
Procedure: hypnosis — It will be proposed to the patient to participate in a study to assess the tolerance of Examination under hypnosis The examination is then conducted in endoscopy room. The patient will benefit from an induction technique of hypnosis by a doctor trained in hypnosis and local anesthesia performed by the endoscopist. In the control group, only local anesthesia is practiced by the endoscopist. The waning, it will ask the patient and endoscopist to complete an evaluation form tolerance of the review
  Arms: Examination under hypnosis in addition to local anesthesia

SUMMARY:
Bronchoscopy is an examination performed routinely in pulmonology. This exam is considered as uncomfortable by nearly 60% of patients, especially due to respiratory blocking sensation, cough and nausea it causes, despite the use of a local anesthetic. Conversely, this examination is rarely performed under general anesthesia in hospitals in France, because it lengthens the duration of the procedure, increases its cost and can be dangerous for the respiratory failure patient.

Hypnosis is an altered state of consciousness between wakefulness and sleep, which can cause the patient to ignore the reality in which he is focusing his attention on his imagination, reducing his anxiety, his painful or unpleasant perceptions and their memorization.

The hypnosis benefit has already been evaluated in the control of pain and anxiety in many medical situations, surgical, obstetric and dental. In endoscopy, the results are mixed. In bronchoscopy, hypnosis has, to our knowledge, not been evaluated.

In a preliminary study in the endoscopy unit of the Hospital Saint Joseph, involving 66 patients, investigators showed that bronchoscopy was poorly tolerated in more than half of patients and that this poor tolerance was correlated to the level anxiety of patients, but 75% of patients surveyed would prefer the waning redo the examination in the same conditions if their health required it, rather than using a general anesthetic. Investigators then hypothesized that hypnosis would improve tolerance bronchoscopy under local anesthesia, without the need for general anesthesia.

DETAILED DESCRIPTION:
Primary objective:

To compare the safety of bronchoscopy performed under local anesthesia and hypnosis to that performed under local anesthesia alone.

Secondary objectives:

* Self-assessment of pain, difficulty breathing, coughing and sensation of nausea experienced by the patient.
* Straight-tolerance assessment of the review by the endoscopist.
* Evaluation of the quality of implementation of the review by the endoscopist.
* Evaluation of the amount of local anesthetic used during the examination.
* Measure the length of the review.

Development of the study:

If the eligibility criteria are present, it will be proposed to the patient to participate in a study to assess the tolerance of Examination under hypnosis. A fact sheet will be handed to him explaining the purpose of the study and the place of examination. If he agrees to participate, consent will be obtained in writing and will be randomized into one of two groups. He will fill a questionnaire clinical information and Anxiety Questionnaire HAD (Hospital Anxiety and Depression Scale). The examination is then conducted in endoscopy room. In the hypnosis group, the patient will benefit from an induction technique of hypnosis by a doctor trained in hypnosis and local anesthesia performed by the endoscopist. In the control group, only local anesthesia is practiced by the endoscopist. The waning, it will ask the patient and endoscopist to complete an evaluation of the tolerance of the examination questionnaire.

Methodology :

DESIGN:

Number of subjects required: 126

The prevalence of poor tolerance of the examination in this population was 52% (numeric scale of the overall tolerance> 3) and the expected objective in the intervention group under hypnosis is a halving of the number of patients with EN > 3 to the overall safety, the number of subjects to be included is 63 per group.

Time study: baseline in January 2015 for an expected period of eight months depending on the pace of inclusion estimated to average 4 per week.

Randomization:

Randomization in the 2 groups will be made by day of the week carries the hypnotherapist (Monday or Tuesday with a random alternation between these 2 days). The list of days will be balanced by randomly alternating blocks. The team of bronchoscopy and prescribers of the bronchoscopy will not be informed of the first schedule to avoid selection bias of patients.

Acquisition of data:

* Gender, age
* respiratory history
* bronchial endoscopy antecedent
* Admission Status (external or hospitalized)
* analgesic and anxiolytic Processing
* Anxiety Questionnaire HAD (Hospital Anxiety and Depression Scale)
* Pre-medication received
* vital parameters before and after the examination: heart rate, oxygen saturation
* Way passage of the endoscope (nose or mouth)
* Time of endoscopy (between the input and the output of the endoscopy suite)
* Quantity Xylocaine used during the exam
* Sampled
* Score cough, pain and overall tolerance of the digital scale review (self-evaluation by the patient)
* Acceptance or not the patient to repeat the examination under the same conditions if his health required in the future
* Straight-evaluation by the physician endoscopist of the overall tolerance of the review by the patient (digital scale)
* Easy to complete the review by the endoscopist (digital scale)
* Summary of potential adverse events

Statistical analysis:

To find and test differences, univariate analyzes will use the test t-Student for continuous variables and the chi of 2 for categorical variables or their nonparametric equivalents. The significance level was set at p <0.05.

1.2 Serious Adverse Event (SAE)

A serious event is an event:

* The evolution of which is fatal; or
* Which endangers the life of the person undergoing research; or
* Which causes a disability or a significant or lasting disability; or
* Causing hospitalization or prolongation of hospitalization; or
* Which results in an abnormality or birth defect; or
* Any other event does not meet the qualifications listed above, but can be regarded as "potentially serious" including some laboratory abnormalities; or
* Medically relevant event in the judgment of the investigator; or
* Events requiring medical intervention to prevent progression to one of the aforementioned states.

The term "life-threatening" is reserved for immediate life-threatening at the time of the adverse event, regardless of the consequences of corrective or palliative therapy.

Certain circumstances requiring hospitalization are not within the gravity standard "inpatient / hospitalization extension" as:

admission for social or administrative reasons; hospitalization predefined by the protocol; hospitalization for medical or surgical treatment scheduled prior research; passing day hospital.

2. detection methods and collection of adverse events:

All adverse events should be investigated, reported and recorded, processed and evaluated the first visit (inclusion Day 0) until the end of the study until their resolution.

Adverse events are collected:

* In clinical, biological and other planned and systematic examination by the investigator;
* By spontaneous reporting by the participants, who will be instructed to contact the investigating doctor in case of adverse events.

All adverse events will be recorded on forms on adverse events of case report form (see Appendix 6). Each observed adverse events will be recorded individually. The intensity of adverse events will be determined as follows:

* Mild (grade 1): no interference on the patient's daily activities;
* Moderate (grade 2): Moderate interference on the patient's daily activities but still acceptable;
* Severe (grade 3) significant interference on the patient's daily activity and unacceptable;
* Threat of life-threatening (grade 4);
* Death (Grade 5). All adverse events must be graded. Responsibilities of the investigator

2.1 Statement of SAEs

The investigator evaluates each adverse event in relation to its severity. The investigator must notify by fax (01 44 12 32 52) to the sponsor (CRC GHPSJ) without delay after the day he heard, all serious adverse events in the trial, except from those identified in the protocol as not requiring immediate reporting. This initial notification is the subject of a written report must be followed if necessary by one or the report (s) Additional (s) writing (s) Main (s) within 8 days of the first declaration.

The investigator must document the best event (thanks to copies of laboratory results or reports of examinations or hospitalization accounts informing the serious event, including relevant negative results, not forgetting to make these documents and anonymous to register number and the patient's code), medical diagnosis and a causal link between serious adverse events and research.

The statement is sent to the developer with the serious adverse event reporting form signed and dated.

The investigator should follow the patient with an SAE to its resolution, stabilization at a level deemed acceptable by the investigator or return to the previous state, even if the patient is out of the test and inform the promoter (CRC GHPSJ) fax: 01 44 12 32 52 using the form (check: monitoring).

2.2 Assessment of causality

The investigator should assess causality of adverse events with research. The causal link is binary (connected / not connected).

2.3 Reporting period and followed the terms of adverse events

The investigator should report serious adverse events from the inclusion of the patient until the end of the experimental procedure.

The investigator should monitor adverse events until resolution or stabilization even if the patient is out of the study.

2.4 Special Cases

2.4.1 Serious Events not immediately declare

To the extent it is expected no serious adverse event related to the participation of patients in this study and that only certain serious adverse events known to be associated with bronchoscopy (hemoptysis, asthma, respiratory distress, allergic xylocaine etc.) may occur, they do not require immediate notification in accordance with the health authorities.

3. Responsibilities of the promoter

The Promoter will declare to ANSM and the CPP in accordance with the law of 9 August 2004:

* all unexpected serious adverse reactions without delay and at the latest within seven calendar days from the day when the sponsor becomes aware of, and within 7 days for monitoring,
* developments without delay safety and at the latest within 7 calendar days, and within 7 days for monitoring,
* annual safety reports within 60 calendar days of the anniversary date of the study.

  4. Appointment of an independent monitoring committee

To the extent it is expected no serious adverse event related to the participation of patients in this study, Investigators do not want to establish an independent monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

* Before performing a bronchoscopy under his medical care
* No opposition to participate in the study

Exclusion Criteria:

* Poor understanding of the French language
* major hearing impairment
* severe cognitive or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-07-04 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety Questionnaire HAD (Hospital Anxiety and Depression Scale) | At Day 0 within 30 minutes after the exam
Assessment of timing change of endoscopy | At Day 0, Time laps Start at the input of the endoscopy suite and stop when the output of the endoscopy suite

CONTACTS AND LOCATIONS:
Overall Officials: Stephane JOUVESHOMME, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France